CLINICAL TRIAL: NCT03663192
Title: Strain Echocardiography During Septic Shock : an Observational Pilot Study
Acronym: Sepsistrain
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB : 16.02.07
Record Dates: First submitted 2018-04-05; First posted 2018-09-10 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2019-05

CONDITIONS: Shock, Septic; Echocardiography
Keywords: Shock, Septic; Echocardiography; speckle tracking; strain
MeSH Terms: conditions — Shock, Septic; Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: strain echocardiography — strain echocardiography during septic shock

SUMMARY:
The mortality of septic shock remains high nowadays despite a trend toward improvement.Septic cardiomyopathy has been reported in most experimental models of sepsis shock. Its relationship with mortality is unclear. A decrease in mortality have been reported in patients with decreased left ventricular ejection fraction (LVEF), but a recent meta-analysis did not support such results. In fact, it appears that high LVEF are linked to profound vasoplegia which is associated to bad outcome.

In the other hand, alterations of Strain echocardiography, a new method allowing a more sensitive evaluation of heart function, have been associated with a worse outcome in sepsis patients. Only few studies have examined echocardiographic strain during sepsis shock in human, and its natural history was only described in pigs. Moreover, the right ventricular strain was reported only by Orde et al whereas the evolution of strain during fluid infusion have never been studied. The aim of the present study is to describe the natural history of echocardiographic strain during sepsis shock and to determine its prognosis value.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock (suspected or proven infection and norepinephrine ≥ 0,25µg/kg/min)
* Inclusion within the first 24h of septic shock

Exclusion Criteria:

* Patient < 18 year of age
* Pregnant women
* History of myocardial infarction, valvular disease, atrial fibrillation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Global peak systolic longitudinal strain assessed by echocardiography. Global peak systolic longitudinal strain | up to 90 days

SECONDARY OUTCOMES:
ICU mortality | up to 90 days
  On the day of patient discharge from the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Claire Roger, MD,PhD, Principal Investigator — CHU Nimes
Locations (1):
- Intensive care unit CHU Nimes, Nîmes, France

REFERENCES:
- [Result] Bazalgette F, Roger C, Louart B, Daurat A, Bobbia X, Lefrant JY, Muller L. Prognostic value and time course evolution left ventricular global longitudinal strain in septic shock: an exploratory prospective study. J Clin Monit Comput. 2021 Dec;35(6):1501-1510. doi: 10.1007/s10877-020-00620-w. Epub 2020 Nov 20. PMID 33216237